CLINICAL TRIAL: NCT00587080
Title: Stapled TransAnal Rectal Resection (STARR): Correlation Between Clinical and Radiological Outcome
Brief Title: Stapled TransAnal Rectal Resection (STARR): Clinical and Radiological Outcome
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Daniel Dindo, MD, University Hospital Zurich
Other Study IDs: StV 33-2006
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Obstructed Defecation Syndrome (ODS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the correlation between clinical and radiological outcome after Stapled TransAnal Rectal Resection (STARR)

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* clinical signs of ODS with prior not effective conservative treatment
* anterior rectoceles and/or intussusceptions in MR-defecography

Exclusion Criteria:

* < 18 years
* fixed enteroceles
* severe fecal incontinence
* external rectal prolapse
* anismus

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ODS and diagnosis of rectal redundancy (intussusception/rectoceles) in MR defecography
Enrollment: 24 (Actual)
Dates: Start 2004-01; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Clinical and radiological outcome as assessed by closed-configuration MR defecography

SECONDARY OUTCOMES:
Morbidity and Mortality after STARR

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dindo, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital, Clinic for Visceral and Transplantation Surgery, Zurich, Canton of Zurich, Switzerland